CLINICAL TRIAL: NCT05660135
Title: Reduction Efficacy of OLOMAX for Blood Pressure and Low-density Lipoprotein Cholesterol in Hypertensive Patients With Dyslipidemia: a Multi-center-database Real-world Study
Brief Title: Reduction Efficacy of OLOMAX for Blood Pressure and Low-density Lipoprotein Cholesterol in Hypertensive Patients With Dyslipidemia
Status: Active, not recruiting | Type: Observational
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Other Study IDs: DWOLM_RWE02
Record Dates: First submitted 2022-12-13; First posted 2022-12-21 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Hypertension; Dyslipidemias
MeSH Terms: conditions — Hypertension; Dyslipidemias | interventions — Olmesartan Medoxomil; Amlodipine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with hypertension and dislipidemia: received olomax tablet as treatment.
  Interventions: Drug: Olmesartan Medoxomil/ Amlodipine Besylate/ Rosuvastatin Ca

INTERVENTIONS:
Drug: Olmesartan Medoxomil/ Amlodipine Besylate/ Rosuvastatin Ca — Olomax Tab 20/5/5mg Olomax Tab 20/5/10mg Olomax Tab 40/5/5mg Olomax Tab 40/5/10mg

SUMMARY:
This study is a large-scale, prospective, multi-center, and non-interventional observation study to observe blood pressure and blood lipid changes and safety during administration of olomax tablets for 24 weeks in hypertensive patients with dyslipidemia.

DETAILED DESCRIPTION:
In this study, investigator will evaluate subjects' clinical performance in actual care. Laboratory test results such as demographic information and medical treatment, blood pressure, blood lipid test, and liver function test conducted at the start date of Olomax tablet administration and subsequent 24 weeks (± 8 weeks) will be collected. In the case of safety-related information, such as abnormal cases, data shall be collected at any time during the 24-week follow-up period if there is a visit by the study subject according to daily treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Adult aged 19 or older at the time of the baseline visit.
2. A patient with hypertension and dyslipidemia who is scheduled to administer olomax tablet according to investigator's medical judgement.

   * Patients who were previously taking more than two tablets of a single drug, low-density lipoprotein-cholesterol (LDL-C)
   * Patients who were previously only taking blood pressure-lowering drugs and did not take LDL-C-lowering drugs, but who need to take additional LDL-C-lowering drugs at the discretion of the researcher
   * Patients who were previously taking LDL-C lowering agents and did not take blood pressure lowering agents, but who need to take additional blood pressure lowering agents according to the researcher's judgment
   * Patients who have not previously taken both a blood pressure drop and an LDL-C drop but need additional simultaneous use at the discretion of the researcher
3. A person who can understand the information provided to him/her and may voluntarily sign a written consent form

Exclusion Criteria:

1. A person who falls under the prohibition of administration according to the permission for olomax tablet
2. A person who has a history of administering olomax tablets before participating in this study
3. In addition to the above, a person that the investigator thinks he/she is not suitable for participating in this observation study;

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is to confirm the effect of olomax tablet -reducing blood pressure and LDL-C- in patients with hypertension and dyslipidemia compared to existing drugs . Of the total 4,672,648 statin prescriptions in 2020, about 295,379 were combined prescriptions for hypertension treatment. It was expected that about 1% of them could be registered, and therefore we estimated 4,000 study subjects to be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2022-06-20 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The rate of change in LDL-C | at 24 weeks
  The rate of change in LDL-C at 12 weeks from baseline
The amount of change in LDL-C | at 24 weeks
  The amount of change in LDL-C at 24 weeks from baseline

SECONDARY OUTCOMES:
The rate of change in LDL-C | at 12 weeks
  The rate of change in LDL-C at 12 weeks from baseline
The amount of change in LDL-C | at 12 weeks
  The amount of change in LDL-C at 12 weeks from baseline
The rate of change in SBP(Systolic Blood Pressure) | 12 weeks
  The rate of change in SBP(Systolic Blood Pressure) at 12 weeks from baseline
The rate of change in SBP(Systolic Blood Pressure) | 24 weeks
  The rate of change in SBP(Systolic Blood Pressure) at 24 weeks from baseline
The amount of change in SBP(Systolic Blood Pressure) | 12 weeks
  The amount of change in SBP(Systolic Blood Pressure) at 12 weeks from baseline
The amount of change in SBP(Systolic Blood Pressure) | 24 weeks
  The amount of change in SBP(Systolic Blood Pressure) at 24 weeks from baseline
The rate of change in lipid variable(TC, HDL-C, non-HDL-C, TG) | 12 weeks
  The rate of change in lipid variable(TC, HDL-C, non-HDL-C, TG) at 12 weeks from baseline
The rate of change in lipid variable(TC, HDL-C, non-HDL-C, TG) | 24 weeks
  The rate of change in lipid variable(TC, HDL-C, non-HDL-C, TG) at 24 weeks from baseline
The amount of change in lipid variable(TC, HDL-C, non-HDL-C, TG) | 12 weeks
  The amount of change in lipid variable(TC, HDL-C, non-HDL-C, TG) at 12 weeks from baseline
The amount of change in lipid variable(TC, HDL-C, non-HDL-C, TG) | 24 weeks
  The amount of change in lipid variable(TC, HDL-C, non-HDL-C, TG) at 24 weeks from baseline
Percentage of subjects who reached LDL-C target | 12 weeks
  Percentage of subjects who reached LDL-C target according to Korean Society of Lipid/Arteriosclerosis's risk classification in the guidelines for the treatment of dyslipidemia (2018) at 12 weeks from baseline
Percentage of subjects who reached LDL-C target | 24 weeks
  Percentage of subjects who reached LDL-C target according to Korean Society of Lipid/Arteriosclerosis's risk classification in the guidelines for the treatment of dyslipidemia (2018) at 24 weeks from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Hun-Sung Kim, Principal Investigator — The Catholic University of Korea
Locations (1):
- The Catholic University of Korea, Seoul ST. Mary's Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
Do not have plan yet